CLINICAL TRIAL: NCT04830969
Title: Impact of Periodontal Therapy on Patients With Diabetes: A Pilot Study
Brief Title: Impact of Periodontal Therapy on Patients With Diabetes
Acronym: DMRCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Sunstar, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Schifferle, DDS, PhD, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000962
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type II; Periodontitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontitis | interventions — Chlorhexidine; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- A: Diabetic + SRP + SPT (Experimental): The first group, A, includes diabetics with periodontal disease; they will receive standard therapy, scaling & root planing plus supportive periodontal therapy (SPT) chlorhexidine gluconate (Paroex®) mouthrinse + Soft-Picks.
  Interventions: Drug: Chlorhexidine gluconate oral rinse; Procedure: Scaling & Root Planing; Device: Soft Picks
- B: Non-Diabetic + SRP + SPT (Experimental): The second group, B, includes non-diabetics with periodontal disease; they will receive standard therapy, scaling & root planing plus supportive periodontal therapy (SPT) chlorhexidine gluconate (Paroex®) mouthrinse + Soft-Picks.
  Interventions: Drug: Chlorhexidine gluconate oral rinse; Procedure: Scaling & Root Planing; Device: Soft Picks
- C: Diabetic + SRP (Active Comparator): The third group, C, includes diabetics with periodontal disease; they will receive standard therapy, scaling and root planing (SRP).
  Interventions: Procedure: Scaling & Root Planing
- D: Non-Diabetic + SRP (Active Comparator): The second group, D, includes non-diabetics with periodontal disease; they will receive standard therapy, scaling and root planing (SRP).
  Interventions: Procedure: Scaling & Root Planing

INTERVENTIONS:
Drug: Chlorhexidine gluconate oral rinse — Paroex® is a non-alcohol chlorhexidine preparation. Participants are to use 15 mL morning and evening for 3 months. With use of chlorhexidine, there is risk of reversible staining of teeth and the possibility of some alteration in taste. There is increased likeliness of staining in smokers, coffee drinkers and those who are susceptible to teeth staining in general. The cleaning of the front teeth is provided at the 3-month visit and helps to reduce any staining that may occur. If there is any alteration in taste, it should go away when use of chlorhexidine stops.
  Other Names: Paroex
  Arms: A: Diabetic + SRP + SPT; B: Non-Diabetic + SRP + SPT
Procedure: Scaling & Root Planing — SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
  Other Names: SRP
Device: Soft Picks — Soft Picks are a rubber interdental bristle cleaner. Participants are to use Soft Picks morning and evening for all 12 months of the study. They may cause some bleeding of the gums at first usage, but the bleeding should lessen and stop as use is continued (as gums heal). Soft-Picks are a readily available consumer product sold in supermarkets and drug stores.
  Arms: A: Diabetic + SRP + SPT; B: Non-Diabetic + SRP + SPT

SUMMARY:
With poorly controlled diabetes, periodontal status often worsens, and with severe periodontal conditions there is often poorer glycemic control. There are few published reports investigating the efficacy of periodontal therapy in diabetics and fewer that include evaluation of the oral microbial profiles (the microbiome). The investigators will examine systemic changes in diabetes status and microbiome influences on clinical response to periodontal therapy in a randomized clinical trial of participants with and without diabetes and with periodontal disease. Two different treatments will be used:

1. Scaling and root planning (SRP) alone, or
2. SRP and supportive periodontal therapy (SPT), the use of chlorhexidine gluconate rinse (Paroex®) and a rubber interdental bristle cleaner (Soft-Picks) The main goal of this clinical trial is to evaluate the effects of SRP alone versus SRP+SPT on clinical, microbiological and immunological status in participants. A clearer understanding of how periodontal therapy affects diabetes status could lead to the development of new therapies for periodontal disease and diabetes.

DETAILED DESCRIPTION:
With poorly controlled diabetes, periodontal disease worsens, and with severe periodontal conditions, there is often poorer glycemic control. Published papers conclude that periodontal treatment leads to a reduction in hemoglobin A1c; however, other studies show limited or no improvement. Some patients do not respond well to professional periodontal therapy, even without diabetes, which could be related to poor oral hygiene and/or host factors including microbial profiles. There are few published papers investigating the efficacy of periodontal therapy in diabetics and fewer that include assessment of the oral microbiome. The investigators will examine systemic changes in diabetes status and microbiome influences on clinical response to periodontal therapy in a randomized clinical trial. It has been shown that chlorhexidine gluconate rinse leads to significant clinical improvement over standard periodontal therapy alone, and interdental tooth cleaners remove more dental plaque (leading to reduced gingival inflammation) effectively than brushing alone. Therefore, in this study, standard periodontal therapy, scaling and root planning (SRP) will be provided alone, or SRP plus supportive periodontal therapy (SPT), the use of chlorhexidine gluconate rinse (Paroex®) and a rubber interdental bristle cleaner (Soft-Picks), to diabetics and non-diabetics with periodontal disease to determine the differences in response between the groups.

The main aim of this study is to evaluate the effects of SRP alone versus SRP+SPT on clinical, microbiological and immunological status of subjects with and without type 2 diabetes and with periodontal disease. A clearer understanding of how periodontal therapy affects diabetes status could lead to the development of novel new targeted therapies of both periodontal disease and diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand the informed consent form and be willing and able to read and sign it.
2. At least 25 years of age.
3. Be able to understand and follow directions for study procedures.
4. At least 14 natural teeth, not counting third molars ("wisdom teeth").
5. At least 2 interproximal sites with CAL >= 4 mm or at least 2 interproximal sites with PD >= 5 mm.

Exclusion Criteria:

1. Presence of orthodontic appliances ("braces").
2. An abnormal condition of lips, lining of the mouth, tongue, or gums (except for periodontal disease). If subject has a cold sore, canker sore, or injury in their mouth, they may return after the sore or injury heals.
3. Abscess of the gingiva caused by periodontal disease, or visible gross tooth decay
4. A broken tooth root or an abscessed tooth. Subject may be allowed to participate in the study after the condition is successfully treated.
5. Periodontal treatment or antibiotic therapy in the past 6 months.
6. Have used cigarettes or other tobacco products in the past year.
7. Body mass index (BMI) is > 40.
8. Have regularly used non-steroidal anti-inflammatory drugs (such as >= 325 mg aspirin or ibuprofen) over the past 3 weeks.
9. Regularly using drugs that weaken the immune system (such as corticosteroids taken by mouth or injection, and cyclosporine).
10. Have participated in another clinical research study in the past 30 days.
11. Pregnant or breastfeeding.
12. Have a condition that we feel will make study participation unsafe or difficult for the patient.
13. Require premedication for dental exams.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Schifferle, DDS, PhD, Principal Investigator — University at Buffalo, State University of New York
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson RG, Shlossman M, Budding LM, Pettitt DJ, Saad MF, Genco RJ, Knowler WC. Periodontal disease and NIDDM in Pima Indians. Diabetes Care. 1990 Aug;13(8):836-40. doi: 10.2337/diacare.13.8.836. PMID 2209317
- [Background] Taylor GW, Burt BA, Becker MP, Genco RJ, Shlossman M, Knowler WC, Pettitt DJ. Non-insulin dependent diabetes mellitus and alveolar bone loss progression over 2 years. J Periodontol. 1998 Jan;69(1):76-83. doi: 10.1902/jop.1998.69.1.76. PMID 9527565
- [Background] Arora N, Papapanou PN, Rosenbaum M, Jacobs DR Jr, Desvarieux M, Demmer RT. Periodontal infection, impaired fasting glucose and impaired glucose tolerance: results from the Continuous National Health and Nutrition Examination Survey 2009-2010. J Clin Periodontol. 2014 Jul;41(7):643-52. doi: 10.1111/jcpe.12258. Epub 2014 May 25. PMID 24708451
- [Background] Engebretson S, Kocher T. Evidence that periodontal treatment improves diabetes outcomes: a systematic review and meta-analysis. J Periodontol. 2013 Apr;84(4 Suppl):S153-69. doi: 10.1902/jop.2013.1340017. PMID 23631575
- [Background] Sgolastra F, Severino M, Pietropaoli D, Gatto R, Monaco A. Effectiveness of periodontal treatment to improve metabolic control in patients with chronic periodontitis and type 2 diabetes: a meta-analysis of randomized clinical trials. J Periodontol. 2013 Jul;84(7):958-73. doi: 10.1902/jop.2012.120377. Epub 2012 Oct 29. PMID 23106512
- [Background] Engebretson SP, Hyman LG, Michalowicz BS, Schoenfeld ER, Gelato MC, Hou W, Seaquist ER, Reddy MS, Lewis CE, Oates TW, Tripathy D, Katancik JA, Orlander PR, Paquette DW, Hanson NQ, Tsai MY. The effect of nonsurgical periodontal therapy on hemoglobin A1c levels in persons with type 2 diabetes and chronic periodontitis: a randomized clinical trial. JAMA. 2013 Dec 18;310(23):2523-32. doi: 10.1001/jama.2013.282431. PMID 24346989
- [Background] Borgnakke WS, Chapple IL, Genco RJ, Armitage G, Bartold PM, D'Aiuto F, Eke PI, Giannobile WV, Kocher T, Kornman KS, Lang NP, Madianos PN, Murakami S, Nishimura F, Offenbacher S, Preshaw PM, Rahman AU, Sanz M, Slots J, Tonetti MS, Van Dyke TE. The multi-center randomized controlled trial (RCT) published by the journal of the American Medical Association (JAMA) on the effect of periodontal therapy on glycated hemoglobin (HbA1c) has fundamental problems. J Evid Based Dent Pract. 2014 Sep;14(3):127-32. doi: 10.1016/j.jebdp.2014.04.017. Epub 2014 May 21. PMID 25234213
- [Background] Colombo AP, Boches SK, Cotton SL, Goodson JM, Kent R, Haffajee AD, Socransky SS, Hasturk H, Van Dyke TE, Dewhirst F, Paster BJ. Comparisons of subgingival microbial profiles of refractory periodontitis, severe periodontitis, and periodontal health using the human oral microbe identification microarray. J Periodontol. 2009 Sep;80(9):1421-32. doi: 10.1902/jop.2009.090185. PMID 19722792
- [Background] Colombo AP, Bennet S, Cotton SL, Goodson JM, Kent R, Haffajee AD, Socransky SS, Hasturk H, Van Dyke TE, Dewhirst FE, Paster BJ. Impact of periodontal therapy on the subgingival microbiota of severe periodontitis: comparison between good responders and individuals with refractory periodontitis using the human oral microbe identification microarray. J Periodontol. 2012 Oct;83(10):1279-87. doi: 10.1902/jop.2012.110566. Epub 2012 Feb 10. PMID 22324467
- [Background] Kirst ME, Li EC, Alfant B, Chi YY, Walker C, Magnusson I, Wang GP. Dysbiosis and alterations in predicted functions of the subgingival microbiome in chronic periodontitis. Appl Environ Microbiol. 2015 Jan;81(2):783-93. doi: 10.1128/AEM.02712-14. Epub 2014 Nov 14. PMID 25398868
- [Background] Wang J, Qi J, Zhao H, He S, Zhang Y, Wei S, Zhao F. Metagenomic sequencing reveals microbiota and its functional potential associated with periodontal disease. Sci Rep. 2013;3:1843. doi: 10.1038/srep01843. PMID 23673380
- [Background] Perez-Chaparro PJ, Goncalves C, Figueiredo LC, Faveri M, Lobao E, Tamashiro N, Duarte P, Feres M. Newly identified pathogens associated with periodontitis: a systematic review. J Dent Res. 2014 Sep;93(9):846-58. doi: 10.1177/0022034514542468. Epub 2014 Jul 29. PMID 25074492
- [Background] Beiswanger BB, Mallat ME, Jackson RD, Mau MS, Farah CF, Bosma ML, Bollmer BW, Hancock EB. Clinical effects of a 0.12% chlorhexidine rinse as an adjunct to scaling and root planing. J Clin Dent. 1992;3(2):33-8. PMID 1524682
- [Background] Faveri M, Gursky LC, Feres M, Shibli JA, Salvador SL, de Figueiredo LC. Scaling and root planing and chlorhexidine mouthrinses in the treatment of chronic periodontitis: a randomized, placebo-controlled clinical trial. J Clin Periodontol. 2006 Nov;33(11):819-28. doi: 10.1111/j.1600-051X.2006.00994.x. Epub 2006 Sep 11. PMID 16965522
- [Background] Abouassi T, Woelber JP, Holst K, Stampf S, Doerfer CE, Hellwig E, Ratka-Kruger P. Clinical efficacy and patients' acceptance of a rubber interdental bristle. A randomized controlled trial. Clin Oral Investig. 2014 Sep;18(7):1873-80. doi: 10.1007/s00784-013-1164-3. Epub 2014 Jan 10. PMID 24407549
- [Background] Santos VR, Lima JA, Miranda TS, Goncalves TE, Figueiredo LC, Faveri M, Duarte PM. Full-mouth disinfection as a therapeutic protocol for type-2 diabetic subjects with chronic periodontitis: twelve-month clinical outcomes: a randomized controlled clinical trial. J Clin Periodontol. 2013 Feb;40(2):155-62. doi: 10.1111/jcpe.12040. PMID 23305133
- [Derived] Li L, Hayashi-Okada Y, Falkner KL, Cervi S, Andrusz S, Shimizu Y, Zambon JJ, Kirkwood KL, Schifferle RE, Diaz PI. Randomized Trial to Test a Chemo-Mechanical Antiplaque Regimen as Adjunct to Periodontal Therapy. JDR Clin Trans Res. 2024 Apr;9(2):160-169. doi: 10.1177/23800844231167065. Epub 2023 May 6. PMID 37148266

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 116 enrolled participants, 114 met inclusion criteria and were randomized for treatment
Groups:
- A: SRP + SPT: The first group, A, includes diabetics and non-diabetics with periodontal disease; they will receive standard therapy, scaling & root planing plus supportive periodontal therapy (SPT) chlorhexidine gluconate (Paroex®) mouthrinse + Soft-Picks.
  Chlorhexidine gluconate oral rinse: Paroex® is a non-alcohol chlorhexidine preparation. Participants are to use 15 mL morning and evening for 3 months. With use of chlorhexidine, there is risk of reversible staining of teeth and the possibility of some alteration in taste. There is increased likeliness of staining in smokers, coffee drinkers and those who are susceptible to teeth staining in general. The cleaning of the front teeth is provided at the 3-month visit and helps to reduce any staining that may occur. If there is any alteration in taste, it should go away when use of chlorhexidine stops.
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
  Soft Picks: Soft Picks are a rubber interdental bristle cleaner. Participants are to use Soft Picks morning and evening for all 12 months of the study. They may cause some bleeding of the gums at first usage, but the bleeding should lessen and stop as use is continued (as gums heal). Soft-Picks are a readily available consumer product sold in supermarkets and drug stores.
- B: SRP: The second group, B, includes diabetics and non-diabetics with periodontal disease; they will receive standard therapy, scaling and root planing (SRP).
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
Period: Overall Study
Arm/Group | A: SRP + SPT | B: SRP
Started | 58 | 56
Completed | 45 | 41
Not Completed | 13 | 15
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Protocol Violation | 3 | 9
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: In this study, unit participant is assigned to Arms/Groups in all measures. For each participant, 6 sites per tooth are evaluated. The measured sites within each participant were summarized to access the outcome in each subject. And the outcome of each participant were analyzed in each Aim.
Groups:
- Diabetic + SRP + SPT: The group includes diabetics with periodontal disease; they will receive standard therapy, scaling & root planing plus supportive periodontal therapy (SPT) chlorhexidine gluconate (Paroex®) mouthrinse + Soft-Picks.
  Chlorhexidine gluconate oral rinse: Paroex® is a non-alcohol chlorhexidine preparation. Participants are to use 15 mL morning and evening for 3 months. With use of chlorhexidine, there is risk of reversible staining of teeth and the possibility of some alteration in taste. There is increased likeliness of staining in smokers, coffee drinkers and those who are susceptible to teeth staining in general. The cleaning of the front teeth is provided at the 3-month visit and helps to reduce any staining that may occur. If there is any alteration in taste, it should go away when use of chlorhexidine stops.
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
  Soft Picks: Soft Picks are a rubber interdental bristle cleaner. Participants are to use Soft Picks morning and evening for all 12 months of the study. They may cause some bleeding of the gums at first usage, but the bleeding should lessen and stop as use is continued (as gums heal). Soft-Picks are a readily available consumer product sold in supermarkets and drug stores.
- Diabetic + SRP: The group includes diabetics with periodontal disease; they will receive standard therapy, scaling and root planing (SRP).
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
- Non-Diabetic + SRP + SPT: The group includes non-diabetics with periodontal disease; they will receive standard therapy, scaling & root planing plus supportive periodontal therapy (SPT) chlorhexidine gluconate (Paroex®) mouthrinse + Soft-Picks.
  Chlorhexidine gluconate oral rinse: Paroex® is a non-alcohol chlorhexidine preparation. Participants are to use 15 mL morning and evening for 3 months. With use of chlorhexidine, there is risk of reversible staining of teeth and the possibility of some alteration in taste. There is increased likeliness of staining in smokers, coffee drinkers and those who are susceptible to teeth staining in general. The cleaning of the front teeth is provided at the 3-month visit and helps to reduce any staining that may occur. If there is any alteration in taste, it should go away when use of chlorhexidine stops.
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
  Soft Picks: Soft Picks are a rubber interdental bristle cleaner. Participants are to use Soft Picks morning and evening for all 12 months of the study. They may cause some bleeding of the gums at first usage, but the bleeding should lessen and stop as use is continued (as gums heal). Soft-Picks are a readily available consumer product sold in supermarkets and drug stores.
- Non-Diabetic + SRP: The group includes non-diabetics with periodontal disease; they will receive standard therapy, scaling and root planing (SRP).
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
- Total: Total of all reporting groups
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP | Total
Number analyzed (Participants) | 21 | 23 | 24 | 18 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.8) | 66 (8.7) | 65.5 (10.9) | 62.3 (7.3) | 63.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 12 | 9 | 32
  Male | 18 | 15 | 12 | 9 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 23 | 24 | 18 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1 | 0 | 2
  African American | 5 | 1 | 1 | 1 | 8
  Caucasian | 15 | 22 | 22 | 17 | 76
Education [Mean (Standard Deviation); unit: year] | 15.6 (2.4) | 16.1 (2.1) | 15.1 (2.3) | 13.8 (1.8) | 15.2 (2.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.5 (5.1) | 32.5 (6.8) | 29.6 (5.6) | 27.7 (4.9) | 30.7 (5.9)
Smoking History [Count of Participants; unit: Participants]
  Never Smoked | 9 | 15 | 13 | 10 | 47
  Former | 11 | 7 | 11 | 8 | 37
  Unknown | 1 | 1 | 0 | 0 | 2
Alcohol Intake [Count of Participants; unit: Participants]
  Never | 0 | 1 | 2 | 1 | 4
  Former | 7 | 8 | 4 | 3 | 22
  Current | 13 | 11 | 17 | 14 | 55
  Unknown | 1 | 3 | 1 | 0 | 5
Whole Mouth Mean Pocket Depth [Mean (Standard Deviation); unit: mm] | 3 (0.5) | 2.7 (0.2) | 2.9 (0.4) | 2.8 (0.3) | 2.8 (0.4)
Whole Mouth Mean Clinical Attachment Loss [Mean (Standard Deviation); unit: mm] — The clinical attachment loss level is defined as the distance from the Cemento-enamel Junction (CEJ) to the free gingival margin, measured with a periodontal probe. Millimeters of recession (loss of attachment) is recorded as a negative number; when the gingival margin is above the CEJ, the measurement (in millimeters) is recorded as positive.
  mm | 3.5 (0.8) | 3.2 (0.7) | 3.3 (0.7) | 3.3 (0.5) | 3.3 (0.7)
% sites with Pocket Depth ≥ 4 mm per participant [Mean (Standard Deviation); unit: % sites with PD >= 4 mm of a participant] — Unit participant instead of site is assigned to arm/group in this measure. Periodontal PD in millimeters was measured with a UNC-15 periodontal probe on 6 sites per tooth. The percentage of sites with Periodontal PD >= 4 mm per participant is accessed, which represents the portion of deep pocket of the participant, indicating the clinical severity.
  % sites with PD >= 4 mm of a participant | 24.9 (15.8) | 18.7 (7.2) | 21.4 (10.6) | 20.2 (10.6) | 21.3 (11.4)
Bleeding on Probing (BOP) Index per participant [Mean (Standard Deviation); unit: BOP index of a participant] — Unit participant instead of site is assigned to arm/group in this measure. 0 is the absence of gingival bleeding, and 1 is the presence of gingival bleeding after probing and measuring for pocket depth. Bleeding on probing index is defined as the percentage of sites with presence of gingival bleeding after probing in a participant. The value of bleeding on probing index ranges from 0 to 100 for each participant. The bleeding on probing index of each participant is accessed and compared between groups.
  BOP index of a participant | 40 (17.2) | 35.9 (13.4) | 34.9 (11.9) | 35.3 (15.3) | 36.5 (14.3)
Plaque Index (PI) per participant [Mean (Standard Deviation); unit: Plaque Index of a participant] — Unit participant instead of site is assigned to arm/group in this measure. Plaque was visually measured on 6 sites per tooth; 0 is the absence of any plaque. 1 is the presence of plaque. For each participant, 6 sites per tooth were evaluated. The Plaque Index (PI) of each participant was defined as the percentage of sites with plaque. The value of PI ranges from 0 to 100 for each participant. And the PI of each participant were analyzed and compared between groups.
  Plaque Index of a participant | 48.0 (16.7) | 47.1 (13.7) | 38.9 (11.5) | 40.3 (14.6) | 43.6 (14.5)
Hemoglobin A1c [Median (Inter-Quartile Range); unit: % of hemoglobin a1c] | 7 [6.4 to 7.9] | 7 [6.5 to 7.7] | 5.5 [5.2 to 5.7] | 5.2 [5.1 to 5.5] | 6 [5.3 to 7]
Fasting Blood Glucose [Median (Inter-Quartile Range); unit: mg/dL] | 129 [110 to 172] | 135 [112.5 to 188.6] | 92 [83 to 97] | 90 [85 to 98] | 107 [88 to 136]
C-reactive Protein (CRP) [Median (Inter-Quartile Range); unit: mg/L] | 2.5 [1.5 to 3.9] | 1.8 [0.6 to 4.7] | 2.2 [1.4 to 5] | 1.2 [0.6 to 2.1] | 1.9 [0.8 to 3.8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Probing Pocket Depth at the 6-month Post-SRP Completed at Baseline
Description: Periodontal PD in millimeters is measured with a UNC-15 periodontal probe on 6 sites per tooth; site status is compared between timepoints measured
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Group A: SRP + SPT: The group includes patients with periodontal disease; they will receive standard therapy, scaling & root planing plus supportive periodontal therapy (SPT) chlorhexidine gluconate (Paroex®) mouthrinse + Soft-Picks.
  Chlorhexidine gluconate oral rinse: Paroex® is a non-alcohol chlorhexidine preparation. Participants are to use 15 mL morning and evening for 3 months. With use of chlorhexidine, there is risk of reversible staining of teeth and the possibility of some alteration in taste. There is increased likeliness of staining in smokers, coffee drinkers and those who are susceptible to teeth staining in general. The cleaning of the front teeth is provided at the 3-month visit and helps to reduce any staining that may occur. If there is any alteration in taste, it should go away when use of chlorhexidine stops.
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
  Soft Picks: Soft Picks are a rubber interdental bristle cleaner. Participants are to use Soft Picks morning and evening for all 12 months of the study. They may cause some bleeding of the gums at first usage, but the bleeding should lessen and stop as use is continued (as gums heal). Soft-Picks are a readily available consumer product sold in supermarkets and drug stores.
- Group B: SRP: The group includes patients with periodontal disease; they will receive standard therapy, scaling and root planing (SRP).
  Scaling & Root Planing: SRP is standard treatment of periodontitis. It involves using a scaler to remover subgingival plaque and other debris in the space between teeth and gums.
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
mm | -0.25 (0.24) | -0.18 (0.2)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Test type: Superiority; p = 0.16, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

2. Secondary Outcome: Change in Probing Pocket Depth at the 3-month Post-SRP Completed at Baseline
Description: as for outcome 1
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
mm | -0.31 (0.27) | -0.21 (0.22)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Test type: Superiority; p = 0.08, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

3. Secondary Outcome: Changes in Clinical Attachment Level at 3, 6 Months After Treatment at Baseline
Description: The distance from the Cemento-enamel Junction (CEJ) to the free gingival margin is measured with a periodontal probe. Millimeters of recession (loss of attachment) is recorded as a negative number; when the gingival margin is above the CEJ, the measurement (in millimeters) is recorded as positive.
Time Frame: Baseline to 3 months;Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
mm
  Baseline to 3-month | -0.1 (0.29) | -0.2 (0.29)
  Baseline to 6-month | -0.1 (0.25) | -0.12 (0.27)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Baseline to 3 months; Test type: Superiority; p = 0.14, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 2: Comparison: Group A: SRP + SPT vs Group B: SRP; Baseline to 6 months; Test type: Superiority; p = 0.8, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

4. Secondary Outcome: Change in % Sites With Probing Pocket Depth >= 4 mm of a Participant at the 3, 6 Months Post-SRP Completed at Baseline
Description: The analysis is based on the measures of each participant. Participant instead of site is used as unite for arm/group. The measure, % sites with probing pocket depth >= 4 mm within each participant, indicates the portion of deep pocket in a participant. Periodontal PD in millimeters is measured with a UNC-15 periodontal probe on 6 sites per tooth; The percentage of sites with Periodontal PD >= 4 mm within each participant was compared between measured time points.
Time Frame: Baseline to 3 months; Baseline to 6 months
Population: For each participant, 6 sites per tooth are evaluated. The measured sites within each participant were summarized to access the outcome in each participant. The analysis is based on participants.
Measure: Mean (Standard Deviation); unit: % sites with PD >= 4 mm of a participant
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
% sites with PD >= 4 mm of a participant
  Baseline to 3-month | -8.71 (7.03) | -4.74 (5.1)
  Baseline to 6-month | -7.03 (6.72) | -4.73 (5.35)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Baseline to 3 months; Test type: Superiority; p < 0.01, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 2: Comparison: Group A: SRP + SPT vs Group B: SRP; Test type: Superiority; p = 0.09, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

5. Secondary Outcome: Changes in Bleeding on Probing (BOP) Index of a Participant at 3, 6 Months After Treatment at Baseline
Description: The analysis is based on the measures of each participant. 0 is the absence of gingival bleeding and 1 is the presence of gingival bleeding after probing and measuring for pocket depth. Bleeding on probing index is defined as the percentage of sites with presence of gingival bleeding after probing per participant. The value of bleeding on probing index ranges from 0 to 100 for each participant. The bleeding on probing index per participant is compared between time points measured.
Time Frame: Baseline to 3 months; Baseline to 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: BOP index of a participant
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
BOP index of a participant
  Baseline to 3 months | -13.24 (9.69) | -5.57 (10.1)
  Baseline to 6 months | -8.93 (10.76) | -4.09 (9.22)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Baseline to 3 months; Test type: Superiority; p < 0.01, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 2: Comparison: Group A: SRP + SPT vs Group B: SRP; Baseline to 6 months; Test type: Superiority; p = 0.03, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

6. Secondary Outcome: Change in Plaque Index of a Participant at 3, 6 Months After Treatment at Baseline
Description: The analysis is based on the measures of each participant. Plaque is visually measured on 6 sites per tooth; 0 is the absence of any plaque. 1 is the presence of plaque. For each participant, 6 sites per tooth are evaluated. The Plaque Index (PI) of each participant is defined as the percentage of sites with plaque. The value of PI ranges from 0 to 100 for each participant. The PI of each participant is assessed and compared between measured time points.
Time Frame: Baseline to 3 months; Baseline to 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Plaque Index of a participant
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
Plaque Index of a participant
  Baseline to 3 months | -14.76 (11.52) | -7.7 (12.5)
  Baseline to 6 months | 9.68 (12.22) | -5.19 (12.08)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Baseline to 3 months; Test type: Superiority; p < 0.01, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 2: Comparison: Group A: SRP + SPT vs Group B: SRP; Baseline to 6 months; Test type: Superiority; p = 0.09, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

7. Secondary Outcome: Change in Probing Pocket Depth at 3, 6 Months After Treatment in Diabetics and Non-diabetics
Description: Probing depth (PD) or probing pocket depth (PPD), measured on six surfaces/tooth, is the distance in millimeters (mm) from the gingival margin to the base of the gingival pocket
Time Frame: Baseline to 3 months; Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
mm
  Baseline to 3-month | -0.36 (0.29) | -0.17 (0.17) | -0.26 (0.24) | -0.27 (0.26)
  Baseline to 6-month | -0.27 (0.27) | -0.12 (0.19) | -0.24 (0.21) | -0.26 (0.19)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.86, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 3: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.047, t-test, 2 sided
Statistical Analysis 4: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.75, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

8. Secondary Outcome: Changes in Clinical Attachment Level at 3, 6 Months After Treatment at Baseline in Diabetics and Non-diabetics
Description: as for outcome 3
Time Frame: Baseline to 3 months; Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
mm
  Baseline to 3 months | -0.11 (0.28) | -0.17 (0.25) | -0.1 (0.31) | -0.23 (0.33)
  Baseline to 6 months | -0.14 (0.24) | -0.06 (0.24) | -0.07 (0.26) | -0.19 (0.29)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.44, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.22, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 3: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.29, t-test, 2 sided
Statistical Analysis 4: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.15, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

9. Secondary Outcome: Change in % Sites With Probing Pocket Depth >= 4 mm of a Participant at the 3, 6 Months Post-SRP Completed at Baseline in Diabetics and Non-diabetics
Description: The analysis is based on the measure of each participant. Periodontal PD in millimeters is measured with a UNC-15 periodontal probe on 6 sites per tooth; The percentage of sites with Periodontal PD >= 4 mm per participant is compared between measured time points.
Time Frame: Baseline to 3 months; Baseline to 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % sites with PD >= 4 mm of a participant
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
% sites with PD >= 4 mm of a participant
  Baseline to 3-month | -10.23 (7.88) | -4.22 (4.22) | -7.39 (6.05) | -5.4 (6.12)
  Baseline to 6-month | -7.85 (8.02) | 4.12 (5.55) | -6.3 (5.41) | -5.52 (5.13)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.31, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 3: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.08, t-test, 2 sided
Statistical Analysis 4: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.54, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

10. Secondary Outcome: Changes in Bleeding on Probing (BOP) Index of a Participant at 3, 6 Months After Treatment at Baseline in Diabetics and Non-diabetics
Description: as for outcome 5
Time Frame: Baseline to 3 months; Baseline to 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: BOP index of a participant
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
BOP index of a participant
  Baseline to 3 months | -13.45 (11.31) | -4.35 (10.62) | -13.06 (8.27) | -7.13 (9.45)
  Baseline to 6 months | -9.62 (13.34) | -1.95 (8.83) | -8.32 (8.12) | -6.82 (9.23)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.04, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 3: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 4: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.38, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

11. Secondary Outcome: Change in Plaque Index of a Participant at 3, 6 Months After Treatment at Baseline in Diabetics and Non-diabetics
Description: as for outcome 6
Time Frame: Baseline to 3 months; Baseline to 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Plaque Index of a participant
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
Plaque Index of a participant
  Baseline to 3 months | -17.46 (13.19) | -7.67 (13.16) | -12.4 (9.48) | -7.75 (11.99)
  Baseline to 6 months | -12.11 (14.05) | -4.97 (12.43) | -7.56 (10.18) | -5.48 (11.96)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.02, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 3 months; Test type: Superiority; p = 0.18, t-test, 2 sided; used generalized linear models adjusted for baseline CRP
Statistical Analysis 3: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.08, t-test, 2 sided
Statistical Analysis 4: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Baseline to 6 months; Test type: Superiority; p = 0.41, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

12. Secondary Outcome: Changes in Hemoglobin A1c at 6 Months After Treatment
Description: Hemoglobin in A1c (HbA1c) tells the average level of blood sugar over the prior 2 to 3 months. Normal level is below 5.7%; 5.7%-6.4% indicates prediabetes; greater than 6.5% is indicative of diabetes.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: % of hemoglobin a1c
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
% of hemoglobin a1c | -0.01 (0.55) | 0.14 (0.72)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Test type: Superiority; p = 0.27, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

13. Secondary Outcome: Changes in Fasting Blood Glucose at 6 Months After Treatment
Description: Fasting blood sugar/glucose (FBS/FBG) is tested with a blood sample taken after an overnight fast. A fasting blood sugar level less than 100 mg/dL is normal; a fasting blood sugar level from 100 to 125 mg/dL is considered prediabetes; a level 126 mg/dL (7 mmol/L) or higher on two separate tests, indicates diabetes.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
mg/dL | -2.13 (32.30) | 1.85 (34.68)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Test type: Superiority; p = 0.54, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

14. Secondary Outcome: Change in High Sensitivity C-reactive Protein at 6 Months After Treatment
Description: The high-sensitivity C-reactive protein (hs-CRP) blood test measures body inflammation indicating infection or a chronic inflammatory disease such as periodontitis or diabetes. It also can be used to evaluate risk of developing coronary artery disease. A normal reading is less than 10 milligram per liter (mg/L); a level greater than 10 mg/L is a sign of serious infection, trauma or chronic disease likely requiring further testing to determine cause
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
mg/L | -0.33 (4.31) | -1.25 (8.84)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Test type: Superiority; p = 0.12, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

15. Secondary Outcome: Changes in Hemoglobin A1c at 6 Months After Treatment in Diabetics and Non-diabetics
Description: as for outcome 12
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: % of hemoglobin a1c
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
% of hemoglobin a1c | -0.04 (0.79) | 0.30 (0.92) | 0.01 (0.18) | -0.07 (0.20)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Test type: Superiority; p = 0.20, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Test type: Superiority; p = 0.07, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

16. Secondary Outcome: Changes in Fasting Blood Glucose at 6 Months After Treatment in Diabetics and Non-diabetics
Description: as for outcome 13
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
mg/dL | -5.05 (46.99) | 2.74 (46.04) | 0.42 (7.78) | 0.72 (9.22)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Test type: Superiority; p = 0.58, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Test type: Superiority; p = 0.64, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

17. Secondary Outcome: Change in High Sensitivity C-reactive Protein at 6 Months After Treatment in Diabetics and Non-diabetics
Description: as for outcome 14
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
Number analyzed (Participants) | 21 | 23 | 24 | 18
mg/L | 0.23 (2.11) | -2.23 (11.82) | -0.41 (5.57) | 0.01 (0.56)
Statistical Analysis 1: Comparison: Diabetic + SRP + SPT vs Diabetic + SRP; Test type: Superiority; p = 0.46, t-test, 2 sided
Statistical Analysis 2: Comparison: Non-Diabetic + SRP + SPT vs Non-Diabetic + SRP; Test type: Superiority; p = 0.11, t-test, 2 sided; used generalized linear models adjusted for baseline CRP

18. Secondary Outcome: Shannon Index of the Subgingival Plaque Microbiome at Baseline and 6 Months
Description: Shannon index represents mean species diversity in a site at a local scale. Shannon index quantifies the uncertainty in predicting the species identity of an individual that is taken at random from the dataset. The minimum value is 0 and there is no maximum value. High values mean high species diversities.
Time Frame: Baseline; 6 Months
Measure: Mean (Standard Deviation); unit: Shannon index value
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
Shannon index value
  Baseline | 5.31 (0.48) | 5.27 (0.55)
  6 Months | 5.2 (0.5) | 5.34 (0.5)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; at baseline; Test type: Superiority; p = 0.7, t-test, 2 sided
Statistical Analysis 2: Comparison: Group A: SRP + SPT vs Group B: SRP; 6 months; Test type: Superiority; p = 0.29, t-test, 2 sided

19. Secondary Outcome: Change in Distance to the Healthy Plane Based on the Subgingival Plaque Microbiome at 6 Months
Description: Analysis of microbiome community changes using the healthy plane (HP) as a reference. A healthy plane was calculated by fitting a plane that minimizes the sum of squares of distances from HC samples to the nearest point on the plane. The distance of each sample to the HP was then calculated. Higher values of distance to HP mean microbiome community changes towards disease status
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: distance to the healthy plane
Arm/Group | Group A: SRP + SPT | Group B: SRP
Number analyzed (Participants) | 45 | 41
distance to the healthy plane | -2.16 (5.84) | -1.26 (7.37)
Statistical Analysis 1: Comparison: Group A: SRP + SPT vs Group B: SRP; Test type: Superiority; p = 0.53, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 Months After Treatment at Baseline
Arm/Group | Diabetic + SRP + SPT | Diabetic + SRP | Non-Diabetic + SRP + SPT | Non-Diabetic + SRP
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23 | 0/24 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 0/24 | 0/18
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 0/24 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04830969/Prot_SAP_000.pdf